CLINICAL TRIAL: NCT04340414
Title: Safety and Effectiveness Study of Low Flow Extracorporeal Membrane Oxygenation（CO2 Removal） Driving by Continuous Hemofiltration Machine the Severe New Corovirus Pneumonia (NCP)
Brief Title: Safety and Effectiveness of Low-flow ECMO Driving by CVVH Machine in Severe NCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Low flow-ECMO by CVVH in NCP
Record Dates: First submitted 2020-03-03; First posted 2020-04-09 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; ECMO
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NCP patient with severe ARDS and/or high ventilator supported (Experimental): The NCP patient with severe ARDS and/or high ventilator supported condition was eligibilitable for enrollment
  Interventions: Device: Low flow ECMO driving by CVVH machine

INTERVENTIONS:
Device: Low flow ECMO driving by CVVH machine — With aim to clear CO2 and improve oxygenation, a low flow ECMO treatment(using oxgyenator membrane of kid type ) driving by CVVH machine will be performed in the NCP with severe ARDS

SUMMARY:
assess the safety and effectiveness of using low-flow extracorporeal membrane oxygenation(CO2 removal) driving by CVVH machine in the severe NCP patients

ELIGIBILITY:
Inclusion Criteria:

* 1. NCP with severe acute respiratory distress syndrome with ratio of partial pressure of arterial oxygen over fraction of inspired oxygen (PaO2:FiO2)<150 and PEEP >10cmH2O
* 2. Driving pressure> 20cmH2O
* 3. RR>30bpm
* 4.PaCO2>55cmH2O and/or PH>7.3

Exclusion Criteria:

* 1. poor venous vascular condition and unavaible for central venous catheter placement

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
PaCO2 | Day 1
  PaCO2 from blood gas analysis
Driving Pressure | Day 1
  Driving Pressure monitor by ventilator
Tidal volume | Day 1
  Tidal volume monitor by ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, Principal Investigator — Peking Union Medical College Hospit
Locations (1):
- Yun Long, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ding X, Chen H, Zhao H, Zhang H, He H, Cheng W, Wang C, Jiang W, Ma J, Qin Y, Liu Z, Wang J, Yan X, Li T, Zhou X, Long Y, Zhang S. ECCO2R in 12 COVID-19 ARDS Patients With Extremely Low Compliance and Refractory Hypercapnia. Front Med (Lausanne). 2021 Jul 8;8:654658. doi: 10.3389/fmed.2021.654658. eCollection 2021. PMID 34307397